CLINICAL TRIAL: NCT05323045
Title: A First-in-human Dose-escalation and Expansion Trial With the Antibody-drug Conjugate BYON3521 to Evaluate the Safety, Pharmacokinetics and Efficacy in Patients With c-MET Expressing Locally Advanced or Metastatic Solid Tumours
Brief Title: A First-in-human Dose-escalation and Expansion Study With the Antibody-drug Conjugate BYON3521
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Byondis B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BYON3521.001
Record Dates: First submitted 2022-03-25; First posted 2022-04-12 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor
Keywords: ADC; c-MET; solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BYON3521 (Experimental): c-MET targeting Antibody-Drug Conjugate
  Interventions: Drug: BYON3521

INTERVENTIONS:
Drug: BYON3521 — BYON3521 (in the vein) infusion every three weeks. Number of cycles: until cancer progression or unacceptable toxicity develops. Different doses.

SUMMARY:
This is the first-in-human trial with BYON3521, an antibody-drug conjugate (ADC) comprising a humanized IgG1 monoclonal antibody directed against the c-MET receptor covalently conjugated to a duocarmycin-containing linker-drug.

DETAILED DESCRIPTION:
This trial includes a dose-escalation part (Part 1) in which the MTD and RDE will be determined, and an expansion part (Part 2) to evaluate efficacy and safety in specific patient cohorts.

BYON3521 is an ADC comprising a humanized IgG1 monoclonal antibody (mAb) directed against the c-MET receptor covalently and site-specifically conjugated to a duocarmycin-containing linkerdrug.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically-confirmed, locally advanced or metastatic cancer who has progressed on standard therapy or for whom no standard therapy exists:
* Part 1 (dose-escalation): solid tumours of any origin;
* Part 2 (expansion):

  * Cohort A: Non-squamous non small cell lung cancer (non-squamous NSCLC);
  * Cohort B: Gynaecological cancers: ovarian cancer, endometrial cancer, cervical cancer;
  * Cohort C: Pancreatic adenocarcinoma (PA);
  * Cohort D: Uveal melanoma (UM).
* c-MET prevalence confirmed by:
* Part 1: Tumour c-MET positive membrane staining by immunohistochemistry (IHC) and/or MET amplification by dual In Situ Hybridization (dISH) and/or known MET-mutation;
* Part 2: Tumour c-MET membrane expression by immunohistochemistry (IHC score ≥ 2+) as determined by the central laboratory on most recent available/obtained tumour material from a site not previously irradiated;
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1;
* Adequate organ function

Exclusion Criteria:

* Having been treated with:
* Trastuzumab duocarmazine (SYD985) at any time;
* Other anticancer therapy within 4 weeks or as defined in the protocol;
* History or presence of keratitis, glomerulonephritis, idiopathic pulmonary fibrosis, organizing pneumonia (e.g. bronchiolitis obliterans), drug-induced or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan;
* History (within 6 months prior to start IMP) or presence of clinically significant cardiovascular disease such as unstable angina, congestive heart failure, myocardial infarction, uncontrolled hypertension, or cardiac arrhythmia requiring medication;
* Symptomatic brain metastases, brain metastases requiring steroids or treatment for brain metastases within 8 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities | 21 days
  Part 1

SECONDARY OUTCOMES:
Objective response rate | 21 days
  Part 2

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Vermaas, Study Director — Byondis B.V., The Netherlands
Locations (4):
- Institut Jules Bordet, Brussels, Belgium
- Istituto Europeo di Oncologia, Milan, Italy
- Radboud, Nijmegen, Netherlands
- Royal Marsden, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Groothuis PG, Jacobs DCH, Hermens IAT, Damming D, Berentsen K, Mattaar-Hepp E, Stokman MEM, Boekel TV, Rouwette M, van der Vleuten MAJ, Sesink A, Dijcks FA, Coumans RGE, Schouten J, Glaudemans DH, Wijk DV, Blomenrohr M, Kappers WA, Ubink R, van der Lee MMC, Dokter WHA. Preclinical Profile of BYON3521 Predicts an Effective and Safe MET Antibody-Drug Conjugate. Mol Cancer Ther. 2023 Jun 1;22(6):765-777. doi: 10.1158/1535-7163.MCT-22-0596. PMID 37042205